CLINICAL TRIAL: NCT02416739
Title: Randomized Double-blinded Comparative Trial to Study the Add-on Activity of Combination Treatment of Nicotinamide on Progression Free Survival for EGFR Mutated Lung Cancer Terminal Stage Patients Being Treated With Gefitinib or Erlotinib
Brief Title: Anticancer Activity of Nicotinamide on Lung Cancer
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Il Yeong Park, Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Il Yeong Park, Ph.D., Professor, Chungbuk National University
Organization: Chungbuk National University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Amina-X-002
Record Dates: First submitted 2015-04-03; First posted 2015-04-15 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Non-Small-Cell Lung Carcinoma
Keywords: EGFR mutated lung cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Niacinamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotinamide (Experimental): Nicotinamide with EGFR-TKI:
  1. gefitinib (250mg tab) or erlotinib (150mg tab) - per oral, once a day
  2. nicotinamide (500mg tab) - per oral, twice a day, until the event or censoring occurs
  Interventions: Drug: Nicotinamide
- Placebo (Placebo Comparator): Placebo tablet with EGFR-TKI:
  1. gefitinib (250mg tab) or erlotinib (150mg tab) - per oral, once a day
  2. placebo tablet - per oral, twice a day, until the event or censoring occurs
  Interventions: Drug: Nicotinamide

INTERVENTIONS:
Drug: Nicotinamide — Nicotinamide (1g/day) or placebo treatment is added to the standard drug treatment (gefitinib or erlotinib) to EGFR mutated NSCLC patients
  Other Names: Amina-X

SUMMARY:
Nicotinamide is an inhibitor of human sirtuins (HDAC III), and is found to re-activate epigenetically silenced tumor suppressors, RUNX3 (runt-related gene 3) and others, in cancer cells. Nicotinamide was found to be effective in several animal cancer models including lung, bladder, liver, etc. The purpose of this study is to determine whether nicotinamide is also effective in the treatment of human lung cancer.

DETAILED DESCRIPTION:
The standard therapy to the EGFR (epidermal growth factor receptor) mutation positive non-small-cell lung cancer patients who are not eligible to operation is to administer EGFR-TKIs (tyrosine kinase inhibitors, gefitinib or erlotinib). To determine the effectiveness of nicotinamide on lung cancer, nicotinamide or placebo tablet will be co-administered with gefitinib or erlotinib for two years until the event or censoring occurs. The stratified block randomization was designed with 3 covariates (EGFR mutation status, kind of EGFR-TKI, ECOG (Eastern Cooperative Oncology Group) performance status score variation). The size of lesions will be checked every other months by radiology. PD (progressive disease) will be assessed according to RECIST(Response Evaluation Criteria in Solid Tumors)1.1. After observing 36 events, an interim analysis of hazard ratio by Cox proportional hazard regression will be performed. The final analysis will be done by the same protocol after observation of 72 events. The significance level of the interim and final analysis were set to 0.0075 and 0.0209 respectively. Response rate, quality of life (measured by 10 questions at every visit), and overall survival will be analysed together. All other adverse reactions will be analysed and reported, if there.

ELIGIBILITY:
Inclusion Criteria:

* Operation-impossible stage 4 non-small-cell lung carcinoma (NSCLC), or recurred terminal stage NSCLC after previous operation or radiation therapy
* EGFR mutated (exon 19 deletion or L858R mutation)
* Life expectation more than 3 months
* More than 1 measurable lesions by RECIST 1.1 which were not exposed to radiation previously
* ECOG (Eastern Cooperative Oncology Group ) performance status grade 0~2
* Who signed the informed consent form

Exclusion Criteria:

* Who had received chemotherapy or EGFR tyrosin kinase inhibitors previously, except whom had received operation at least 6 months ago and received supplementary chemotherapy
* Who has metastasized brain lesion that needs operation or radiation therapy
* Above grade 2, CTCAE (Common Toxicity Criteria for Adverse Effects) 4.0 criteria for blood, liver and kidney
* Who does Not agree to contraception
* Who has allergy to nicotinamide

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Hazard ratio (PFS) of the nicotinamide arm to the placebo arm | two year
  Cox regression analysis

SECONDARY OUTCOMES:
Response rate | two year
  chi-square test of complete response and partial response (RECIST 1.1)
Difference in quality of life between the nicotinamide arm and the placebo arm | two year
  measured by the cancer-related QOL questionaire response (questioned at each visit)
Overall survival | two year
  Cox regression analysis

CONTACTS AND LOCATIONS:
Overall Officials: Il Yeong Park, PhD, Study Director — Chungbuk National University
Locations (1):
- Chonnam National University Hwasun Hospital, Hwasun, Chonnam, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li QL, Kim HR, Kim WJ, Choi JK, Lee YH, Kim HM, Li LS, Kim H, Chang J, Ito Y, Youl Lee K, Bae SC. Transcriptional silencing of the RUNX3 gene by CpG hypermethylation is associated with lung cancer. Biochem Biophys Res Commun. 2004 Jan 30;314(1):223-8. doi: 10.1016/j.bbrc.2003.12.079. PMID 14715269
- [Background] Li QL, Ito K, Sakakura C, Fukamachi H, Inoue Ki, Chi XZ, Lee KY, Nomura S, Lee CW, Han SB, Kim HM, Kim WJ, Yamamoto H, Yamashita N, Yano T, Ikeda T, Itohara S, Inazawa J, Abe T, Hagiwara A, Yamagishi H, Ooe A, Kaneda A, Sugimura T, Ushijima T, Bae SC, Ito Y. Causal relationship between the loss of RUNX3 expression and gastric cancer. Cell. 2002 Apr 5;109(1):113-24. doi: 10.1016/s0092-8674(02)00690-6. PMID 11955451
- [Background] Avalos JL, Bever KM, Wolberger C. Mechanism of sirtuin inhibition by nicotinamide: altering the NAD(+) cosubstrate specificity of a Sir2 enzyme. Mol Cell. 2005 Mar 18;17(6):855-68. doi: 10.1016/j.molcel.2005.02.022. PMID 15780941
- [Background] Black JC, Mosley A, Kitada T, Washburn M, Carey M. The SIRT2 deacetylase regulates autoacetylation of p300. Mol Cell. 2008 Nov 7;32(3):449-55. doi: 10.1016/j.molcel.2008.09.018. PMID 18995842
- [Background] Lee YS, Lee JW, Jang JW, Chi XZ, Kim JH, Li YH, Kim MK, Kim DM, Choi BS, Kim EG, Chung JH, Lee OJ, Lee YM, Suh JW, Chuang LS, Ito Y, Bae SC. Runx3 inactivation is a crucial early event in the development of lung adenocarcinoma. Cancer Cell. 2013 Nov 11;24(5):603-16. doi: 10.1016/j.ccr.2013.10.003. PMID 24229708
- [Background] Omar MF, Ito K, Nga ME, Soo R, Peh BK, Ismail TM, Thakkar B, Soong R, Ito Y, Salto-Tellez M. RUNX3 downregulation in human lung adenocarcinoma is independent of p53, EGFR or KRAS status. Pathol Oncol Res. 2012 Oct;18(4):783-92. doi: 10.1007/s12253-011-9485-5. Epub 2012 Jun 24. PMID 22729835
- [Background] Kim WJ, Lee JW, Quan C, Youn HJ, Kim HM, Bae SC. Nicotinamide inhibits growth of carcinogen induced mouse bladder tumor and human bladder tumor xenograft through up-regulation of RUNX3 and p300. J Urol. 2011 Jun;185(6):2366-75. doi: 10.1016/j.juro.2011.02.017. Epub 2011 Apr 21. PMID 21511279
- [Background] Park SY, Lee KB, Lee MJ, Bae SC, Jang JJ. Nicotinamide inhibits the early stage of carcinogen-induced hepatocarcinogenesis in mice and suppresses human hepatocellular carcinoma cell growth. J Cell Physiol. 2012 Mar;227(3):899-908. doi: 10.1002/jcp.22799. PMID 21503886
- [Background] Surjana D, Halliday GM, Damian DL. Role of nicotinamide in DNA damage, mutagenesis, and DNA repair. J Nucleic Acids. 2010 Jul 25;2010:157591. doi: 10.4061/2010/157591. PMID 20725615
- [Background] Peck B, Chen CY, Ho KK, Di Fruscia P, Myatt SS, Coombes RC, Fuchter MJ, Hsiao CD, Lam EW. SIRT inhibitors induce cell death and p53 acetylation through targeting both SIRT1 and SIRT2. Mol Cancer Ther. 2010 Apr;9(4):844-55. doi: 10.1158/1535-7163.MCT-09-0971. Epub 2010 Apr 6. PMID 20371709
- [Background] McCarthy AR, Sachweh MC, Higgins M, Campbell J, Drummond CJ, van Leeuwen IM, Pirrie L, Ladds MJ, Westwood NJ, Lain S. Tenovin-D3, a novel small-molecule inhibitor of sirtuin SirT2, increases p21 (CDKN1A) expression in a p53-independent manner. Mol Cancer Ther. 2013 Apr;12(4):352-60. doi: 10.1158/1535-7163.MCT-12-0900. Epub 2013 Jan 15. PMID 23322738
- [Background] Knip M, Douek IF, Moore WP, Gillmor HA, McLean AE, Bingley PJ, Gale EA; European Nicotinamide Diabetes Intervention Trial Group. Safety of high-dose nicotinamide: a review. Diabetologia. 2000 Nov;43(11):1337-45. doi: 10.1007/s001250051536. PMID 11126400
- [Background] Gale EA, Bingley PJ, Emmett CL, Collier T; European Nicotinamide Diabetes Intervention Trial (ENDIT) Group. European Nicotinamide Diabetes Intervention Trial (ENDIT): a randomised controlled trial of intervention before the onset of type 1 diabetes. Lancet. 2004 Mar 20;363(9413):925-31. doi: 10.1016/S0140-6736(04)15786-3. PMID 15043959
- [Background] Petley A, Macklin B, Renwick AG, Wilkin TJ. The pharmacokinetics of nicotinamide in humans and rodents. Diabetes. 1995 Feb;44(2):152-5. doi: 10.2337/diab.44.2.152. PMID 7859933
- [Background] Schoenfeld DA. Sample-size formula for the proportional-hazards regression model. Biometrics. 1983 Jun;39(2):499-503. PMID 6354290
- [Background] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Background] Zhou C, Wu YL, Chen G, Feng J, Liu XQ, Wang C, Zhang S, Wang J, Zhou S, Ren S, Lu S, Zhang L, Hu C, Hu C, Luo Y, Chen L, Ye M, Huang J, Zhi X, Zhang Y, Xiu Q, Ma J, Zhang L, You C. Erlotinib versus chemotherapy as first-line treatment for patients with advanced EGFR mutation-positive non-small-cell lung cancer (OPTIMAL, CTONG-0802): a multicentre, open-label, randomised, phase 3 study. Lancet Oncol. 2011 Aug;12(8):735-42. doi: 10.1016/S1470-2045(11)70184-X. Epub 2011 Jul 23. PMID 21783417
- [Derived] Oh HJ, Bae SC, Oh IJ, Park CK, Jung KM, Kim DM, Lee JW, Kang CK, Park IY, Kim YC. Nicotinamide in Combination with EGFR-TKIs for the Treatment of Stage IV Lung Adenocarcinoma with EGFR Mutations: A Randomized Double-Blind (Phase IIb) Trial. Clin Cancer Res. 2024 Apr 15;30(8):1478-1487. doi: 10.1158/1078-0432.CCR-23-3059. PMID 38593249